CLINICAL TRIAL: NCT06236568
Title: Impact of Graft Reconditioning With Hypothermic Machine Perfusion on HCC Recurrence After Liver Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Paolo Magistri, Assistant Professor of Surgery, Azienda Ospedaliero-Universitaria di Modena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 561/2023/SPER/AOUMO.
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma; Liver Transplant; Complications
Keywords: Hepatocellular carcinoma; Liver Transplantation; Metabolomics; Liquid biopsy; Machine perfusion; Ischemia reperfusion injury
MeSH Terms: conditions — Carcinoma, Hepatocellular; Reperfusion Injury | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Machine perfusion (Experimental): The liver graft to be transplanted is treated with 90 minutes of D-HOPE machine perfusion
  Interventions: Device: D-HOPE machine perfusion; Procedure: Liver transplantation
- No machine perfusion (Active Comparator): Standard liver transplantation
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Device: D-HOPE machine perfusion — use of the device
  Arms: Machine perfusion
Procedure: Liver transplantation — Liver transplantation for HCC within Milan criteria

SUMMARY:
The use of devices for liver grafts perfusion before transplantation, either hypothermic (HOPE) or normothermic (NMP), is rapidly spreading thanks to the promising results obtained so far in terms of graft survival and post-operative morbidity. Besides the well-established ability to increase the rate of transplantability of extended criteria donors (ECD) and donors after cardiac death (DCD), the use of machine perfusion (MP) may also improve the oncological outcomes of patients affected by hepatocellular carcinoma (HCC) undergoing liver transplantation (LT). The underlying mechanism is represented by the modulation of the ischemia-reperfusion injury (IRI)-related cellular damage obtained by the liver graft perfusion with HOPE before LT. The identification of biomarkers able to predict graft outcomes and highlight the mechanism of graft injury before transplantation rapidly and in non-invasive manner is therefore needed. Mass spectrometry-based metabolomics has already shown its potential by using perfusion liquids or pre-implantation biopsies.

The aim of the investigators is to run an open-label, randomised, controlled trial to study the impact of treating standard liver grafts from brain dead donors (DBD) with HOPE before liver transplant in patients affected by HCC. Patients aged 18-75 years presenting with HCC Milan-in at listing will be considered for inclusion. Presence of extra-hepatic disease and general contraindications to liver transplantation as defined by the local tumor board are considered as exclusion criteria. Eligible patients will be randomly assigned (1:1) with the use of a dedicated software to MP (intervention group) or no-MP (control group) before liver transplantation. Untargeted mass spectrometry metabolomics (UHPLC-HRMS) will be performed on liver graft perfusate, liver graft biopsy and recipient blood samples, to identify by classification methods, novel predictive markers of IRI. Furthermore, rapid targeted MS approaches will be performed on VIP metabolites and known key compounds (such as TCA, aminoacids, energy metabolism) to rapidly assess graft function as well as post-operative outcome.

Blood samples of the recipient will be collected at two checkpoints (listing, and 3 months after liver transplant) to evaluate exosomes and miRNA expression fluctuations (liquid biopsy).

Primary outcomes of the study will be overall survival, graft survival and recurrence-free survival at 1- and 2-years. Survival results will be compared to those expected based on the Metroticket 2.0 score to assess the impact of MP in reducing the risk of HCC recurrence. Patients will remain in follow-up as for clinical practice to assess 3- and 5-years survival. Secondary end-point will be to define liquid biopsy efficacy to predict HCC recurrence and to define the correlation between metabolomic observations and HCC recurrence pattern.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCC within Milan criteria at listing candidate for liver transplantation
* ECOG 0-2
* DBD donors
* capability to sign an informed consent

Exclusion Criteria:

* pediatric patients
* DCD donors
* DBD extended criteria requiring machine perfusion (no ethical randomization)
* living donor liver transplantation
* split liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 5 years after surgery
  Recurrence free survival and overall survival after LT for HCC according to the use of MP This aim will be realized at the Hepato-pancreato-biliary Surgery and Liver Transplantation Unit of Policlinico University Hospital of Modena - University of Modena and Reggio Emilia, supervised by Dr Paolo Magistri. Patients included in the trial according to the following criteria will be treated and followed-up according to the standard of care (SOC). All eligible patients have an indication to LT beyond the aims of this study, and will undergo LT according to National indications. LT is the gold standard treatment for patients affected by HCC inside Milan criteria, however biological features of the tumor may modify the expected recurrence pattern.
  This aim will be focused on the potential role for MP in the modulation of tumor recurrence pattern.
  SA1 Deliverables:
  Modulation of HCC recurrence pattern after MP

SECONDARY OUTCOMES:
Prognostic markers - MiRNA | 5 years after surgery
  Identification of microRNAs from liquid biopsy derived extracellular vesicles, as source of prognostic information on IRI favoring HCC recurrence. This aim will be realized by Research Laboratory at Policlinico University Hospital of Modena - University of Modena and Reggio Emilia, supervised by Dr Valentina Masciale.
  SA2 Deliverables:
  1) miRNAs transcriptomic profile of pre transplanted-patients.
Prognostic markers - metabolipiodomics | 5 years after surgery
  Identification of at least 1 prognostic markers from the promising miRNA selected on the bases of the transcriptomic analysis.
  SA3: Identification of prognostic markers of IRI and HCC by MS-based metabolipidomics:
  This aim will be realized by UNIT2, Unisa-Difarma, Dr. Eduardo Maria Sommella
Graft survival | 1 month after surgery
  Reduction of early allograft disfunction

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Di Benedetto, Study Chair — University of Modena and Reggio Emilia; Massimo Dominici, Study Chair — University of Modena and Reggio Emilia; Pietro Campiglia, Study Chair — University of Salerno; Eduardo M Sommella, Principal Investigator — University of Salerno; Valentina Masciale, Principal Investigator — University of Modena and Reggio Emilia; Ilenia Mastrolia, Principal Investigator — University of Modena and Reggio Emilia
Locations (1):
- AOU di Modena, Modena, MO, Italy

IPD SHARING:
Plan to Share IPD: Undecided